CLINICAL TRIAL: NCT03177460
Title: A Pilot Presurgical Study of Daratumumab (CD38 Antagonist) or JNJ-40346527 in Men With High-Risk Localized Prostate Cancer Followed by Radical Prostatectomy
Brief Title: Daratumumab or FMS Inhibitor JNJ-40346527 Before Surgery in Treating Patients With High-Risk, Resectable Localized or Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0103; NCI-2018-01179 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0103 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Prostate Adenocarcinoma; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Testosterone Greater Than 150 ng/dL
MeSH Terms: conditions — Prostatic Neoplasms | interventions — daratumumab; JNJ-40346527

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (daratumumab) (Experimental): Patients receive daratumumab IV over 4-8 hours once weekly for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo radical prostatectomy during week 6.
  Interventions: Biological: Daratumumab; Procedure: Radical Prostatectomy
- Arm B (FMS inhibitor JNJ-40346527) (Experimental): Patients receive FMS inhibitor JNJ-40346527 PO BID for 4-5 weeks in the absence of disease progression or unacceptable toxicity. After a 3 day wash-out period, patients undergo radical prostatectomy.
  Interventions: Drug: FMS Inhibitor JNJ-40346527; Procedure: Radical Prostatectomy

INTERVENTIONS:
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
  Arms: Arm A (daratumumab)
Drug: FMS Inhibitor JNJ-40346527 — Given PO
  Other Names: JNJ-40346527
  Arms: Arm B (FMS inhibitor JNJ-40346527)
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy

SUMMARY:
This phase I trial studies the side effects of daratumumab or FMS inhibitor JNJ-40346527 before surgery in treating patients with high-risk prostate cancer that can be removed by surgery and has not spread to other parts of the body or has spread to nearby tissue or lymph nodes. Immunotherapy with monoclonal antibodies, such as daratumumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spreadFMS inhibitor JNJ-40346527 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving daratumumab or FMS inhibitor JNJ-40346527 before surgery may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Safety and tolerability of therapy with the study drugs in men with high-risk localized prostate cancer.

SECONDARY OBJECTIVES:

I. To assess the proportion of patients who achieve pathological complete response (CR) with the study drugs in men with high-risk localized prostate cancer.

EXPLORATORY OBJECTIVES:

I. To study immunological changes in tumor tissues and peripheral blood in response to the study drugs in men with high-risk localized prostate cancer.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM A: Patients receive daratumumab intravenously (IV) over 4-8 hours once weekly for 4 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo radical prostatectomy during week 6.

ARM B: Patients receive FMS inhibitor JNJ-40346527 orally (PO) twice daily (BID) for 4-5 weeks in the absence of disease progression or unacceptable toxicity. After a 3 day wash-out period, patients undergo radical prostatectomy.

After completion of study treatment, patients are followed up at week 18.

ELIGIBILITY:
Inclusion Criteria:

* Consent to MD Anderson laboratory protocol PA13-0291.
* Histological documentation of adenocarcinoma of the prostate reviewed at MD Anderson Cancer Center. Patients with small cell, neuroendocrine, or transitional cell carcinomas are not eligible.
* Patients with high-risk prostate cancer (at least 1 core with Gleason sum >= 8) must have at least three core biopsies involved with cancer (a minimum of 6 core biopsies, must be obtained at baseline). A prostate biopsy within 3 months from screening is allowed for entry requirements.
* No evidence of metastatic disease as documented by technetium-99m (99mTc) bone scan and by computed tomography (CT) or magnetic resonance imaging (MRI) scans.
* Eugonadal state (serum testosterone > 150 ng/dL).
* Localized or locally advanced disease deemed by the surgeon to be resectable. Patients must be appropriate candidates for radical prostatectomy plus pelvic lymph node dissection.
* No prior treatment for prostate cancer including prior surgery (excluding transurethral resection of the prostate [TURP]), cryoablation, pelvic lymph node dissection, radiation therapy, hormonal therapy or chemotherapy.
* To avoid risk of drug exposure through the ejaculate (even men with vasectomies), subjects must use a condom during sexual activity while on study drug and for 3 months following the last dose of study drug. If the subject is engaged in sexual activity with a woman of childbearing potential, a condom is required along with another effective contraceptive method consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies and their partners. Donation of sperm is not allowed while on study drug and for 3 months following the last dose of study drug.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) grade of 0 or 1.
* AT SCREENING: Hemoglobin within institutional normal limits. Administration of growth factors or blood transfusions will not be allowed to confirm eligibility.
* AT SCREENING: Platelet count within institutional normal limits. Administration of growth factors or blood transfusions will not be allowed to confirm eligibility.
* AT SCREENING: Absolute neutrophil count within institutional normal limits. Administration of growth factors or blood transfusions will not be allowed to confirm eligibility.
* AT SCREENING: Absolute lymphocyte count within institutional normal limits. Administration of growth factors or blood transfusions will not be allowed to confirm eligibility.
* AT SCREENING: Serum chemistries, renal and liver panels within institutional normal limits or meets the requirements for radical prostatectomy.
* Each subject must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

* Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens, ketoconazole, or estrogens (5-alpha reductase inhibitors allowed), or luteinizing hormone-releasing hormone (LHRH) agonists/antagonists.
* Currently enrolled in another interventional study.
* Concurrent treatment with systemic corticosteroids (prednisone dose > 10 mg per day or equivalent) or other immunosuppressive drugs < 14 days prior to treatment initiation. Steroids that are topical, inhaled, nasal (spray), or ophthalmic solution are permitted.
* History of or known or suspected autoimmune disease (exception[s]: subjects with vitiligo, resolved childhood atopic dermatitis, hypothyroidism, or hyperthyroidism that is clinically euthyroid at screening are allowed).
* Known evidence of an active infection requiring systemic therapy such as human immunodeficiency virus (HIV), active hepatitis, or fungal infection.
* History of clinically significant cardiovascular disease including, but not limited to:

  * Myocardial infarction or unstable angina =< 6 months prior to treatment initiation.
  * Clinically significant cardiac arrhythmia.
  * Deep vein thrombosis, pulmonary embolism, stroke =< 6 months prior to treatment initiation.
  * Congestive heart failure (New York Heart Association class III-IV).
  * Pericarditis/clinically significant pericardial effusion.
  * Myocarditis.
  * Endocarditis.
* History of major implant(s) or device(s), including but not limited to:

  * Prosthetic heart valve(s).
  * Artificial joints and prosthetics placed =< 12 months prior to treatment initiation.
  * Current or prior history of infection or other clinically significant adverse event associated with an exogenous implant or device that cannot be removed.
* Other prior malignancy (exceptions: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) =< 2 years prior to enrollment.
* Any medical, psychological or social condition that in the opinion of the investigator, would preclude participation in this study.
* DARATUMUMAB ONLY: Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [antiHBc] and/or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (antiHBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV deoxyribonucleic acid (DNA) by PCR. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to week 18
  Will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Will be recorded for all patients, recording name, grade, start and end dates, attribution to study drug, and whether the event was alleviated or controlled with relevant appropriate care similar to Phase I trials.

SECONDARY OUTCOMES:
Pathological complete response (CR) | Up to week 18
  Pathologic response will be measured from the surgical specimen. Pathologic CR is defined as the absence of residual tumor in the radical prostatectomy specimen (i.e., pT0).
Immune changes in blood | Baseline up to week 18
Immune changes in tumor tissue | Baseline up to week 18

CONTACTS AND LOCATIONS:
Overall Officials: Sumit K Subudhi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org